CLINICAL TRIAL: NCT02887898
Title: Efficacy of Advanced Carbohydrate Counting and Automated Bolus Calculation in Insulin-treated Type 2 Diabetes Patients: The BolusCal2 Study
Brief Title: Efficacy of Automated Bolus Calculation in Type 2 Diabetes
Acronym: BolusCal2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Merete Bechmann Christensen, MD, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BolusCal2
Record Dates: First submitted 2016-08-15; First posted 2016-09-02 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carb counting and bolus calculator (Active Comparator): Education in carb counting and the use of an automated bolus calculator
  Interventions: Device: Automated bolus calculator; Other: Education
- Carb counting (Placebo Comparator): Education in carb counting and manual calculation of insulin bolus
  Interventions: Other: Education

INTERVENTIONS:
Device: Automated bolus calculator
  Arms: Carb counting and bolus calculator
Other: Education

SUMMARY:
The investigators hypothesize that non-optimal basal-bolus insulin treated patients with type 2 diabetes can achieve better metabolic control by counting carbohydrates with concurrent use of an automated bolus calculator. Additionally, the investigators propose that this intervention will lead to improvement in patient related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes > 1 year
* Age 18 years or older
* HbA1C > 64 mmol/mol (8.0 %)
* Treatment with multiple daily insulin injections (basal and prandial insulin) ≥ 6 months
* GAD-antibody negative
* Naïve to bolus calculators

Exclusion Criteria:

* Pregnancy or breast feeding
* Gastroparesis
* Severe nephropathy (eGFR<30 mL/min/1,73 m2)
* Use of sulfonylurea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | 6 months

SECONDARY OUTCOMES:
Time spent below, in or above the glucose target 4-10 mmol/l measured by continuous glucose monitoring (CGM) | 6 months
Frequency of blood glucose measurements assessed by meter download before randomization and at each visit | 6 months
Frequency of hypoglycemia (below 2.8 mmol/L or unconsciousness/ need of medical assistance) | 6 months
Change in diet habits/diet composition | 6 months
  Assessed by electronic diet recordings
Change in treatment satisfaction | 6 months
  Using questionnaire

OTHER OUTCOMES:
Adherences to bolus calculator use | 6 months
  Using questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark

REFERENCES:
- [Derived] Christensen MB, Serifovski N, Herz AMH, Schmidt S, Hommel E, Raimond L, Perrild H, Gotfredsen A, Gaede P, Norgaard K. Efficacy of Bolus Calculation and Advanced Carbohydrate Counting in Type 2 Diabetes: A Randomized Clinical Trial. Diabetes Technol Ther. 2021 Feb;23(2):95-103. doi: 10.1089/dia.2020.0276. Epub 2020 Sep 21. PMID 32846108